CLINICAL TRIAL: NCT02607202
Title: A Phase II, Randomized, Multicenter Study to Assess the Efficacy of Nab-paclitaxel-based Doublet as First Line Therapy in Patients With Cancer of Unknown Primary (CUP): The AGNOSTOS Trial
Brief Title: A Study of Nab-paclitaxel-based Doublet as First Line Therapy in Patients With Cancer of Unknown Primary (CUP)
Acronym: AGNOSTOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione del Piemonte per l'Oncologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 008-IRCC-10IIS-14
Record Dates: First submitted 2015-11-16; First posted 2015-11-17 (Estimated); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Unknown Primary Tumors
MeSH Terms: conditions — Neoplasms, Unknown Primary | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): nab-paclitaxel 125 mg/m2 on Days 1 and 8 by IV administration over 30 minutes without premedication, followed by gemcitabine 1000 mg/m2 on Days 1 and 8 by IV administration over 30 minutes. Treatment to be repeated Q21 days.
  Interventions: Drug: nab-paclitaxel; Drug: Gemcitabine
- Arm B (Experimental): nab-paclitaxel 125 mg/m2 on Days 1 and 8 by IV administration over 30 minutes without premedication, followed by carboplatin AUC 2 on Day 1 and 8 by IV administration over 60 minutes. Treatment to be repeated Q21 days.
  Interventions: Drug: nab-paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: nab-paclitaxel
  Other Names: Abraxane
Drug: Carboplatin
  Arms: Arm B
Drug: Gemcitabine
  Arms: Arm A

SUMMARY:
Agnostos Trial is a multicentric phase 2 randomized trial with a 'pick-the-winner design' in chemonaive patients with cancer of unknown primary. It will assess the efficacy of the two best active single agent - carboplatin or gemcitabine - added to an innovative taxane back bone (nab-Paclitaxel). Agnostos trial is a part of a larger clinical and translational initiative to improve the outlook of patients with cancer of unknown primary through evaluation of novel chemotherapeutic regimens.

DETAILED DESCRIPTION:
Treatment-naïve patients with CUP diagnosis confirmed according to CUP Diagnostic Guidelines, will be enrolled into AGNOSTOS trial. Patients will be randomized upfront to receive a nab-paclitaxel-based duplet adding either carboplatin or gemcitabine until progression or unacceptable toxicity (randomization 1:1, n= 120; 60 per arm).

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent.
* Patients must be ≥ 18 years of age.
* Diagnosis of CUP according to CUP Diagnostic Guidelines derived from ESMO 2011 and NCCN 2015 guidelines.
* Sufficient archived biopsy tissue from a surgical or core needle biopsy required to perform the CUP multiplex assay.
* Eastern Cooperative Oncology Group performance status ≤ 2.
* No previous systemic therapy.
* At least one measurable lesion by RECIST Criteria.
* Good liver, cardiac, lung and marrow bone function.
* Evidence of non-childbearing status for female patients: negative urine or serum pregnancy test within 21 days of study treatment for women of childbearing potential, or postmenopausal status.
* Patients of child bearing potential and their partners, who are sexually active, must agree to the use of highly effective forms of contraception throughout their participation in the study.
* Patient is willing and able to comply with the protocol for the duration of the study, including undergoing treatment and scheduled visits and examinations.

Exclusion Criteria:

* Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, breast Ductal Carcinoma in Situ (DCIS), stage 1 grade 1 endometrial carcinoma.
* Specific treatable CUP syndromes including: extragonadal germ cell syndrome; neuroendocrine carcinoma; adenocarcinoma isolated to axillary lymph nodes (women cancer); peritoneal carcinomatosis (women - ovarian cancer); squamous carcinoma limited to cervical, supraclavicular, or inguinal lymph nodes; single resectable metastasis.
* Patients receiving any radiotherapy (except for palliative reasons), within 2 weeks from the last dose prior to study entry.
* Patients with symptomatic uncontrolled brain metastases.
* Major surgery within 2 weeks of starting the study and patients must have recovered from any effects of any major surgery.
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 6 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent.
* Pregnant or breast feeding women.
* Immunocompromised patients, eg, patients who are known to be serologically positive for human immunodeficiency virus (HIV).
* Patients with known hepatic disease (eg, Hepatitis B or C).
* Previous cancer treatment.
* Patients currently enrolled in another clinical tria, except AGNOSTOS PROFILING.
* Patients that are receiving chemotherapy, hormonal therapy (HRT is acceptable) or other novel agents.
* Patients receiving live virus and bacterial vaccines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-03; Primary Completion 2021-05-04 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) as evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 guidelines. | 42 months

SECONDARY OUTCOMES:
duration of response according to RECIST version 1.1. | 42 months
time to progression | 42 months
overall survival | 42 months
toxicity according to Common Terminology Criteria for Adverse Events - CTCAE version 4.03. | 42 months

CONTACTS AND LOCATIONS:
Locations (10):
- Italy (10):
  - Investigative Clinical Oncology (Oncologia Medica 2), Candiolo, Turin
  - AOU Policlinoco S Orsola - Malpighi, Bologna
  - Ospedali Galliera, Genova
  - Istituto Europeo di Oncologia - IEO, Milan
  - Istituto Nazionale dei Tumori, Milan
  - Ospedale Niguarda Cà Granda, Milan
  - Istituto Oncologico Veneto - IOV, Padua
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Policlinico Universitario Campus Biomedico, Roma
  - A.O.U S.Giovanni Battista, Torino